CLINICAL TRIAL: NCT02553408
Title: Patients and Care Providers Perspectives and Experience With Decision Aid Tool for Self-monitoring of Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Stewart Harris, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Canada-IIS_ADC-OUS-IIS-14-07
Record Dates: First submitted 2015-09-03; First posted 2015-09-17 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neo meter (Other): This is a single arm purely qualitative (interview only) study with no comparator. All participants will use the FreeStyle Precision Neo-Meter for at least 3 months for self-monitoring of their blood glucose.
  Interventions: Device: FreeStyle Precision Neo-Meter

INTERVENTIONS:
Device: FreeStyle Precision Neo-Meter — Participants will receive a free glucose meter (Neo) and test strips from their care providers with education and instructions on how to use the meter to monitor their glucose level. Three months after the start of using the meter, participants will be interviewed on their experiences, likes and dislikes about the meter.

SUMMARY:
Putting the limited use of titration algorithms in the context of escalating diabetes prevalence rates, strategies and tools are urgently needed to help both patients and primary care providers efficiently initiate and continue basal insulin therapy. Basel insulin is considered to be the appropriate strategy after oral diabetic agent failure. This project could set the stage for the need for a blood glucose meter with built-in algorithms designed to support decision making by patients as well as care providers. Furthermore, the project will evaluate the uptake and use of the newly developed Meter by Abbott Diabetes Care, which was launched in Canada in October 2014, and its impact on primary care diabetes consultation.

DETAILED DESCRIPTION:
The objectives of this study are to

1. Describe patients' and care providers' satisfaction associated with the use of the FreeStyle Precision Neo-Meter
2. Evaluate the uptake and use of the Meter
3. Describe the impact of the Meter on primary care diabetes consultation from care providers' perspectives.

In order to achieve the objectives of this study, diabetes healthcare providers and people with type 2 diabetes who have been using the Neo meter will be interviewed. Maximum variability will be sought for provider discipline and patient demographic characteristics. Sampling will continue until theme saturation is reached. A total of up to 20 (10 care providers and 10 people with diabetes) will be interviewed for this study.

Diabetes healthcare provider interview: Two care providers from each discipline including physicians, nurses, nurse educators and dietitians in Southwestern Ontario, Canada, who have been using the Neo meter will be recruited for interviews. Care providers satisfaction will be assessed after the use of the Meter with sample representation of sole and team based practices.

Patient interviews: Eligible patients who agreed to participate in the study will be provided with a Neo meter and test strips. Their care providers will provide them with instructions, guidance and support in using the device as part of their self-management activities. Patients will be interviewed 3 months after (post only) the use of the Meter to assess their satisfaction with its functionality, capacity, design and ease-of-use.

Interviews will take place at a location and time convenient for participants and will take approximately 45min-60min in Oct/Nov 2015. Interviews will be audio tape recorded to allow for a fluid discussion such that the interviewer does not need to stop the conversation to take notes. A letter of information and consent form will be provided to participants.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with type 2 diabetes and starting basal insulin
* Inadequately managed patients i.e. patients who require further insulin intensification
* Patients who have used the Meter for at least 3 months
* Individuals who are over the age of 17

Exclusion Criteria:

* Individuals with type 1 diabetes
* Individuals who are over the age of 80
* Patients with psychological disorder
* Refuse to use the Meter to test their blood sugar

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Patient and Care provider satisfaction structured interview guide | 3 months after the use of the meter
  Patients and Care providers will be interviewed to assess their satisfaction associated with the use of the meter and its perceived impact on diabetes management.Results will be reported in a qualitative way with participants quotes and themes that will be emerged from the interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Harris, MD, Principal Investigator — The Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No